CLINICAL TRIAL: NCT05975931
Title: A Single-centre, Non-interventional, Retrospective Study to Describe the IMPACT of AspireSR® for Vagus Nerve Stimulation (VNS) Therapy on Healthcare Resource Utilisation and Clinical Outcomes.
Brief Title: IMPACT of AspireSR® for VNS Therapy on Healthcare Resource Utilisation and Clinical Outcomes.
Acronym: IMPACT
Status: Terminated | Type: Observational
Why Stopped: The decision to terminate was taken based on study team capacity not sufficient and alignment with the sponsor.
Sponsor: LivaNova (Industry)
Collaborators: OPEN VIE Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: LNE802
Record Dates: First submitted 2023-07-03; First posted 2023-08-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
Keywords: VNS; Drug Resistant Epilepsy; Vagus Nerve Stimulation; AspireSR®; Health Care Utilization; DRE
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 ("new insertions cohort"): Subjects who have had Aspire SR® implanted as their first VNS model.
- Cohort 2 ("battery change cohort"): Subjects who have had their VNS battery changed from a previous model to Aspire SR®.

SUMMARY:
This is a retrospective non-interventional study to describe the HCRU and clinical outcomes before and after AspireSR® device implantation in subjects with drug resistant epilepsy at the Queen Elizabeth Hospital, Birmingham (QEHB).

DETAILED DESCRIPTION:
Real-world data on healthcare resource use (HCRU) for subjects with treatment-resistant epilepsy and their clinical outcome prior to- and post-VNS device implantation in the UK are limited.

The current study aims to describe and compare the secondary HCRU and clinical outcomes prior to and following AspireSR® device implantation in subjects with drug resistant epilepsy.

Retrospectively-collected data from hospital medical records (paper-based and/or electronic, as appropriate) will be used to describe subject characteristics, disease control and clinical outcomes. All secondary HCRU data will be extracted from the Hospital Episode Statistics (HES) database by Harvey Walsh Ltd (HW, trading under OPEN VIE). Primary HCRU data will be requested from the subjects' general practitioners (GPs).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at AspireSR® device implantation.
* VNS device AspireSR® implantation for the first time or battery change from a previous model to AspireSR® at least 24 months prior to the start of retrospective data collection from medical records.
* Subjects for whom written informed consent has been provided for researcher access to their medical records and extraction of data from HES (if the subject is living and has capacity to consent) or advice from a consultee (if the subject is living but lacks capacity to consent).
* Subjects with available medical history for at least 24 months prior to Aspire SR® implantation.

Exclusion Criteria:

* Living subjects for whom consent for researcher access to medical records and extraction of data from HES has not been obtained.
* Deceased subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult (aged ≥18 years at AspireSR® implantation) subjects with epilepsy who have had the VNS device AspireSR® implanted at least 24 months prior to study retrospective data collection.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Descriptive comparison of healthcare resource use (HCRU) | 24 months before and after device implantation
  Descriptive comparison of secondary HCRU in the 24 month periods before and after AspireSR® device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wysota, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital Birmingham, Birmingham, United Kingdom